CLINICAL TRIAL: NCT00954265
Title: Phase III Study on the Effects of Recombinant HCG Ovulation Triggering on Stimulation, Embryonic and Pregnancy Parameters in an IVF Program
Brief Title: Pregnancy Rates in IVF After Ovulation Triggering With Recombinant or Urinary Human Chorionic Gonadotrophin (HCG)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Dr Papanikolaou Evangelos, Centre for Reproductive Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rec-HCG 002
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-08

CONDITIONS: Embryonic Development; Pregnancy; VEGF
Keywords: pregnancy occurence; OHSS
MeSH Terms: interventions — Chorionic Gonadotropin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Urinary-HCG group (Active Comparator): These patients received u-HCG for ovulation triggering during ovarian stimulation for IVF
  Interventions: Drug: 10000 IU urinary HCG
- Recombinant HCG group (Experimental): These patients received rec-HCG for ovulation triggering during ovarian stimulation for IVF
  Interventions: Drug: 250 mcg recombinant HCG

INTERVENTIONS:
Drug: 10000 IU urinary HCG — ovulation triggering
  Arms: Urinary-HCG group
Drug: 250 mcg recombinant HCG — ovulation triggering
  Arms: Recombinant HCG group

SUMMARY:
To access whether the ovulation triggering with rec-HCG instead urinary-HCG has any impact on the blastulation rate and pregnancy rate of patients undergoing IVF treatment

ELIGIBILITY:
Inclusion Criteria:

* FSH<12,
* normal sperm,less than 36y,
* single blastocyst transfer

Exclusion Criteria:

* endometriosis stage 3&4,
* pco

Ages: 20 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2005-08; Primary Completion 2007-12 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
blastulation rate | on day-5

SECONDARY OUTCOMES:
pregnancy rates, VEGF levels, OHSS rate | 14 days after oocyte pick up

CONTACTS AND LOCATIONS:
Overall Officials: Paul Devroey, Professor, Study Director — Professor or OB-GYN
Locations (1):
- Centre for Reproductive Medicine, UZ Brussel, Brussels, Jette, Belgium